CLINICAL TRIAL: NCT06363032
Title: Application of Transthoracic Shear-wave Ultrasound Elastography in the Evaluation of Renal Function and Diagnosis of Renal Disease
Brief Title: Elastography in Predicting Renal Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202110104RINB
Record Dates: First submitted 2021-12-28; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-12

CONDITIONS: Kidney Disease
Keywords: elastography
MeSH Terms: conditions — Kidney Diseases | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: elastography — When routine renal ultrasound is arranged, patients will be invited to receive elastography at the same time.

SUMMARY:
There are two types of elastography: strain elastography assesses the degree of strain when applying a given amount of force to the skin. Shear-wave elastography assesses the velocity of shear wave propagation within the target lesion. A part of the tissue is deformed by a "push pulse", the velocity of the shear waves propagating within the tissue is detected, and the stiffness of the tissue is assessed based on the detected shear velocity. Shear-wave elastography has been intensively studied in thyroid, breast, liver, cervical lymph nodes, and musculoskeletal diseases with promising result.

Transthoracic shear-wave ultrasound is also used for the prediction of lung malignancy.

In progressive renal disease, renal function decline correlates with the extent of interstitial fibrosis, irrespective of the original pathology. Experience and research in using shear-wave elastography to study the stiffness of renal parenchyma and renal fibrosis are scanty. The investigators will conduct a prospective observational study. This study aims to provide the information of tissue elasticity in different etiologies of renal diseases and to validate the predictive value of shear-wave elastography in predicting renal function and renal fibrosis.

By assuming a power of 0.8, a two-side p value of 0.05, a ratio of 0.2 (sample sizes in negative/positive groups) to detect the difference between area under ROC curve and null hypothesis value (0.8 and 0.7), a target sample of 273 (with a 5% cushion, 260~290) patients is required.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving scheduled renal biopsy and scheduled renal sonography

Exclusion Criteria:

* age < 20 y/o, patients who can't hold their breath for at least 5 seconds

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients receiving scheduled renal biopsy and scheduled renal sonography
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
collect medical record of blood urea nitrogen and Creatinine | 3 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan